CLINICAL TRIAL: NCT01011244
Title: A Phase II Clinical Study of ADIPOPLUS (Autologous Cultured Adipose-derived Stem Cell) for the Treatment of Crohn's Fistula to Evaluate Safety and Efficacy
Brief Title: Safety and Efficacy Study of Autologous Cultured Adipose -Derived Stem Cells for the Crohn's Fistula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTG-ASC-202
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADIPOPLUS (Experimental): patients with a fistula in Crohn's disease
  Interventions: Biological: ADIPOPLUS

INTERVENTIONS:
Biological: ADIPOPLUS — autologous cultured adipose-derived stem cells
  1x10e7 cells/1cm2 depending on surface area of fistula
  Other Names: ANTG-ASC

SUMMARY:
Up to date, a sure cure for Crohn's fistula does not known and the fistula recurrence rate is high. On 15 October 2008, orphan designation was granted by Korea FDA for human adipose-derived stem cell (ADIPOPLUS) for the treatment of Crohn's fistula. In this study, patients are given injection of ADIPOPLUS in fistula site and followed for 8 weeks to evaluate the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Prior diagnosis of Crohn's disease
* patients who have Crohn's fistula
* negative for serum beta-HCG for woman of childbearing age
* agreement to participate, with signed informed-consent

Exclusion Criteria:

* patients who have allergy to bovine-derived materials or an anesthetic
* patients with a diagnosis of auto immune disease except for Crohn's disease
* Diagnosis of HBV, HCV, HIV and other infectious disease
* Patients who have a symptom of septicemia
* Patients with a diagnosis of active Tuberculosis
* Patient who are pregnant or breast-feeding
* Patients who are unwilling to use an "effective" method of contraception during the study
* Patients with a diagnosis of Inflammatory Bowel Disease except for Crohn's disease
* Patients who are sensitive to Fibrin glue
* Patients who have a clinically relevant history of abuse of alcohol or drugs, habitual smoker
* Insufficient adipose tissue for manufacturing of ADIPOPLUS
* Patients who are considered not suitable for the study by investigator
* Patients with a diagnosis of active refractory Crohn's disease
* Patients who have history of surgery for malignant cancer in the past 5 years
* Patients who have > 2 cm diameter of fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy: complete closure of fistula at week 8 | 8 weeks
number of patients with any adverse event | Day 0, Week 8

SECONDARY OUTCOMES:
Photo of target fistula | 8 weeks
  taking Photo of target fistula : Day 0, week 4, 6, 8
number of patients with any adverse events | 8 weeks
  Adverse reaction : day 0, Week 4, 6, 8
number of patients with complete closure of fistula | 8 weeks
  complete closure : every visits more than 50% closure of fistula : every visits
Investigator's satisfaction | 8 weeks
  Investigator's satisfaction : week 8

CONTACTS AND LOCATIONS:
Overall Officials: CS Yu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea